CLINICAL TRIAL: NCT06376305
Title: EndoBarrier Obstructive Sleep Apnoea Study
Brief Title: EndoBarrier in Obstructive Sleep Apnoea Study
Acronym: End-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Bob Ryder (Other)
Collaborators: Association of British Clinical Diabetologists (Unknown)
Responsible Party: Sponsor-Investigator, Dr Bob Ryder, Doctor, Sandwell & West Birmingham Hospitals NHS Trust
Organization: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 176786
Record Dates: First submitted 2024-04-05; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; Obstructive Sleep Apnoea; Obesity
Keywords: EndoBarrier
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EndoBarrier in diabetes with obstructive sleep apnoea (Other): The arm will consist of patients diabetes or prediabetes who also have moderate obstructive sleep apnoea requiring continuous positive pressure ventilation
  Interventions: Device: EndoBarrier

INTERVENTIONS:
Device: EndoBarrier — During screening visit, a brief history, examination, blood tests and 2 sleep studies within a gap of 1 week will be performed. Then, there will be an assessment by gastroenterologist for EndoBarrier insertion. EndoBarrier will be inserted endoscopically as a day case procedure after the midnight fast, under general anaesthesia. Following the EndoBarrier insertion, there will be 3 monthly trial visits until one year where the following assessments will be performed - brief interview, observations, blood tests, urine test, dietitian review, compliance check with CPAP and quality of life questionnaire.
  At the end of one year, EndoBarrier will be removed endoscopically again as a day case procedure under general anaesthesia. Then, there will be follow up trial visits every 3 months up to one year where there will be clinical assessments, sleep studies, blood tests, urine test, dietitian, compliance check and quality of life questionnaires.

SUMMARY:
Obstructive sleep apnoea (OSA) is a common condition in which the upper airways (windpipe) collapse repeatedly during sleep, blocking the flow of air into the lungs. It is characterized by repetitive pauses in breathing during sleep, despite the effort to breathe, and is associated with a reduction in the amount of oxygen in the blood (oxygen saturation). People with OSA are at risk of heart disease, high blood pressure, stroke, depression, and premature death. OSA is usually treated using a continuous positive airway pressure (CPAP) machine. This involves the patient wearing a face mask during sleep which is connected to the machine which supplies a constant steam of air to help keep the airways open. This improves the symptoms and hopefully the long-term outlook, but it is an uncomfortable solution. OSA is associated with obesity and weight loss can improve or even cure it. Treatment with EndoBarrier (placement of a thin flexible tube that is placed inside your intestine creating a physical barrier between the intestinal wall and the food so less can be absorbed) can be associated with significant weight loss and can improve blood sugar control in patients with type 2 diabetes related to their weight (diabesity). This study aims to find out if EndoBarrier treatment can improve OSA in patients with diabesity to the extent that some patients no longer require their CPAP machine treatment.

DETAILED DESCRIPTION:
Once the participant has decided to take part in the study, they will be invited for signing a consent form and screening checks which will include medical history, examination, blood tests (approximately 10 ml) and sleep studies (at home without CPAP) on two occasions within one week to determine whether they are eligible for the study. If they fulfil all the criteria and once recruited into the study, they will be assessed for placement of EndoBarrier by gastroenterologists (tummy doctors) followed by its insertion in City Hospital as a day case procedure. There may be individual or group information sessions including the use of models and videos to describe insertion and removal of EndoBarrier devices. Potential participants will be offered the opportunity to ask questions. There will be trial assessment visits for every 3 months until one year after the insertion of EndoBarrier and then for every 3 months up to one year following its removal. During these visits, participants are assessed clinically and have blood tests (approximately 10 ml taken in a fasted state), sleep studies and quality of life questionnaires. EndoBarrier will be removed after 1 year, again, as a day case procedure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate OSA on CPAP fulfilling NICE criteria for CPAP(AHI between 15 and 29 with symptoms)
* Prediabetes(HbA1c between 42 & 48 mmol/mol) or confirmed type 2 diabetes (HbA1C≥48mmol/mol)
* Obesity BMI ≥30 and ≤45 Kg/m2
* Age ≥ 18 years
* Capable of giving informed consent

Exclusion Criteria:

* Abnormal intestinal anatomy
* Contraindication to oesophagogastroduoenoscopy
* Previous bariatric surgery or bowel surgery
* Active infection
* Anticoagulation therapy
* Coagulopathy INR >1.3
* Estimated Glomerular Filtration Rate (eGFR)<30
* Known portal hypertension
* Uncontrolled cardiovascular disease
* Lactating or pregnant females
* Excess anaesthetic risk
* Patients taking non-steroidal anti-inflammatory agents will need to discontinue these for the duration of Endobarrier implantation
* Patients taking aspirin/clopidogrel with active ischaemic heart disease or cerebrovascular disease(secondary prevention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Requirement for continuous positive airway pressure (CPAP) treatment will be assessed by sleep studies at screening and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Requirement for continuous positive airway pressure

SECONDARY OUTCOMES:
Apnea-hypopnea index (AHI) is measured by sleep studies at screening and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Apnea-hypopnea index (AHI)
Obstructive sleep apnoea (OSA) symptoms are measured by sleep studies at screening, and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Obstructive sleep apnoea (OSA) symptoms
Continuous positive airway pressure (CPAP) pressures are measured by sleep studies at screening, and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Continuous positive airway pressure (CPAP) pressures
Glycated haemoglobin measured by blood test (HbA1c) at screening, baseline, and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Glycated haemoglobin
Fasting plasma glucose is measured by blood test(fasting plasma glucose) at baseline, and then at 12 and 24 months | At baseline, and then at 12 and 24 months
  Fasting plasma glucose
Weight and Body mass index (BMI) is measured by checking weight in kilograms as well as height (in metres) ( weight and height will be combined to report BMI in kg/m^2) at screening, baseline, and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Weight and Body mass index (BMI)
Composite scores of NAFLD severity derived from the blood measurements of Alanine Aminotransferase in U/L, Aspartate Aminotransferase in U/L, platelets in x10^9/L and serum albumin in g/L as well as age in years and BMI | At screening, baseline, and then every 3 months, up to 24 months
  Composite scores of NAFLD severity
Circulating free testosterone, fasting insulin and C-Peptide are measured by blood tests at baseline, and then at 3, 12 and 24 months | At baseline, and then at 3, 12 and 24 months
  Circulating free testosterone, fasting insulin and C-Peptide
Blood pressure is measured by checking blood pressure at sitting at screening, baseline, and then every 3 months, up to 24 months | Every 3 months, up to 24 months
  Blood pressure
Diabetes treatment including need for insulin is measured at baseline, and then every 3 months, up to 24 months21 and 24 months | Every 3 months, up to 24 months
  Diabetes treatment
Quality of life scores is measured by EQ-5D questionnaire at baseline and then at 6, 12 and 24 months | At baseline and then at 6, 12 and 24 months
  Quality of life score

CONTACTS AND LOCATIONS:
Locations (1):
- City Hospital, Birmingham, United Kingdom

REFERENCES:
- [Result] de Jonge C, Rensen SS, Verdam FJ, Vincent RP, Bloom SR, Buurman WA, le Roux CW, Schaper NC, Bouvy ND, Greve JW. Endoscopic duodenal-jejunal bypass liner rapidly improves type 2 diabetes. Obes Surg. 2013 Sep;23(9):1354-60. doi: 10.1007/s11695-013-0921-3. PMID 23526068
- [Result] Schouten R, Rijs CS, Bouvy ND, Hameeteman W, Koek GH, Janssen IM, Greve JW. A multicenter, randomized efficacy study of the EndoBarrier Gastrointestinal Liner for presurgical weight loss prior to bariatric surgery. Ann Surg. 2010 Feb;251(2):236-43. doi: 10.1097/SLA.0b013e3181bdfbff. PMID 19858703